CLINICAL TRIAL: NCT01302704
Title: The Influence of Proton Pump Inhibitors (PPI's) on Blood Levels of 25-Hydroxyvitamin D.
Status: Withdrawn | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20110003H
Record Dates: First submitted 2011-02-17; First posted 2011-02-24 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Vitamin D
Keywords: Vitamin D; Proton Pump Inhibitors

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to demonstrate if Proton Pump Inhibitors (PPI's) decrease blood levels of 25-Hydroxyvitamin D (25-OH Vitamin D).

DETAILED DESCRIPTION:
Subjects (DoD beneficiaries) will be recruited from all male and female subjects whom are at least 18 years of age and are Nellis Air Force Base dependents or retirees. A total of 65 subjects will be recruited.

Screening Visit:

* Obtain signed Informed Consent document and HIPAA Authorization
* Women of child bearing potential will have a serum pregnancy test (approximately 1-2 teaspoons of blood)
* 25-OH Vitamin D baseline levels will be drawn via 1 venipuncture (approximately 1-2 teaspoons of blood)

Visit 1 (within 1 week of screening visit):

• Subjects will be prescribed oral omeprazole 20mg (a proton pump inhibitor) by one of the Investigators. Subject will take oral omeprazole 20mg for 60 consecutive days.

Telephone Call 1 (2 weeks after visit 1):

• Review with the patient (see attached telephone call script)

* If they have been taking the omeprazole 20 mg as prescribed? (studies have shown that patient recall is as accurate as pill counts)
* Review any adverse effects the patient may have experienced.

Telephone Call 2 (2 weeks after Telephone Call 1):

• Review with the patient (see attached telephone call script)

* If they have been taking the omeprazole 20 mg as prescribed? (studies have shown that patient recall is as accurate as pill counts)
* Review any adverse effects the patient may have experienced.

Telephone Call 3 (2 weeks after Telephone Call 2):

* Review with the patient (see attached telephone call script)

  * If they have been taking the omeprazole 20 mg as prescribed? (studies have shown that patient recall is as accurate as pill counts)
  * Review any adverse effects the patient may have experienced.
* Schedule for Final Visit 2.

Final Visit 2 (after 60 days of taking omeprazole):

* Review with the patient:

  * If they have been taking the omeprazole 20 mg as prescribed? (studies have shown that patient recall is as accurate as pill counts)
  * Review any adverse effects the patient may have experienced.
* 25-OH Vitamin D levels will be drawn via 1 venipuncture (approximately 1-2 teaspoons of blood) (research-driven).

Patient's participation in this study is completed after Final Visit 2.

The data will be analyzed and a paper will be written and submitted to a scientific journal.

If at any time during the study, the subject decides to withdraw from the study, they may do so with no further testing required. If a subject becomes pregnant during the study, they will be told to stop omeprazole and withdrawn from the study and referred to their PCM for standard of care treatment.

Patients must agree to take precautions to prevent pregnancy during the course of this study due to the possible severe harm the Omeprazole may cause an unborn child. The only completely reliable methods of birth control are total abstinence or surgical removal of the uterus. Other methods, such as the use of condoms, a diaphragm or cervical cap, birth control pills, IUD, or sperm killing products are not totally effective in preventing pregnancy. Also, women who are breastfeeding may not participate in this study.

If at any time, 25-OH Vitamin D levels are measured and found to be below 10, the patient will be notified immediately to stop taking the oral Omeprazole 20mg and will be referred to their PCM to initiate standard of care treatment.

Oral omeprazole 20mg is a Food & Drug Administration approved dosage. Its use in this protocol is not considered standard of care since it is being used on healthy subjects.

"In accordance with 21 CFR 312.2(b)(i-v), an IND exemption is requested based on the following provisions: (i) The investigation is not intended to be reported to FDA as a well-controlled study in support of a new indication for use nor intended to be used to support any other significant change in the labeling for the drug; (ii) If the drug that is undergoing investigation is lawfully marketed as a prescription drug product, the investigation is not intended to support a significant change in the advertising for the product; (iii) The investigation does not involve a route of administration or dosage level or use in a patient population or other factor that significantly increases the risks (or decreases the acceptability of the risks) associated with the use of the drug product; (iv) The investigation is conducted in compliance with the requirements for institutional review set forth in part 56 and with the requirements for informed consent set forth in part 50; and (v) The investigation is conducted in compliance with the requirements of §312.7."

ELIGIBILITY:
Inclusion Criteria:

* Tricare Insurance Beneficiary (military insurance) receiving care at Nellis AFB
* Male and Female (DoD beneficiaries) at least 18 years of age and have lived in the Las Vegas area for at least 3 months.

Exclusion Criteria:

* Subjects less than 18 years of age.
* Subjects that have known malabsorption conditions.
* 25-OH Vitamin D less than 10
* Pregnancy
* Non English speaking
* Taking any prescription medication or over the counter antacids
* Vitamin d supplements (excluding multivitamin supplements due to relatively low dose of vitamin D)
* Any medical condition that requires regular monitoring by health care provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting healthy volunteers (DoD beneficiaries) whom are at least 18 years of age from the Nellis Air Force Base population. Subjects will not have any concomitant medical conditions, been diagnosed with any chronic illness that requires regular monitoring by a health care provider, have been living in Las Vegas for at least 3 months, and not be on any medications. Some subjects may be the PI or AI's patients. No special populations will be recruited.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in 25-OH Vitamin D Blood Levels over 60 days | 2 years
  Subjects will have their baseline 25-OH Vitamin D levels drawn. They will then take Omeprazole 20mg for 60 consecutive days, then have blood samples drawn to measure their 25-OH Vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Piepenbrink, D.O., Principal Investigator — Michael O'Callaghan Federal Hospital/Nellis Air Force Base
Locations (1):
- Mike O'Callaghan Federal Hospital, Nellis Air Force Base, Nevada, United States